CLINICAL TRIAL: NCT04017676
Title: Optimizing the Resources of Psychotherapy as a Tool for Implementing the Mental Health Reform: A Multicenter Controlled Clinical Trial
Brief Title: Optimizing the Resources of Psychotherapy as a Tool for Implementing the Mental Health Reform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Geha Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sha0006-19
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Psychotherapy Research and Outcome Measures

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, controlled study with a group comparison and a program trial, in which the subjects are recruited according to a systematic allocation by order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The first group will be under the usual treatment conditions (TAU)
- Experimental group (Experimental): The second group will be exposed to a multidisciplinary therapeutic program that has a monitoring component and after two months an intervening component will be.
  Interventions: Other: Supervision assissted by measures

INTERVENTIONS:
Other: Supervision assissted by measures — In the weeks 10 and 13, about 72 hours after the meeting scheduled for that week, and before the next therapeutic session, there will be a structured training session (based on the recommendations of Krägeloh et al., 2015), based on information in the literature about the various questionnaires
  Arms: Experimental group

SUMMARY:
Psychotherapy is one of the cornerstones in public and private mental health services. Despite the tremendous investment in psychotherapy, its efficiency ranges from 40% to 60%. Given the Mental health Reform (2015), aimed at increasing the quality, availability, and accessibility of mental health services, there is an urgent need to manage and maximize psychotherapy services in Israel.

DETAILED DESCRIPTION:
Objectives: To examine the feasibility of implementing managing (monitor and interventional) procedures in psychotherapy services conducted in public mental health services, to assess their effect on the outcome, and to estimate their impact on the 2015 Mental Health Reform objectives.

Working hypotheses:

* After appropriate preparation, managed psychotherapeutic service will be implemented in 4 public mental health out-patients clinics;
* Managed psychotherapeutic service will lead to an improvement in the outcome of psychotherapy;
* Managed psychotherapeutic service will increase the efficacy of mental health services.

Methods:

Type of study: A multicenter, randomized, controlled study with a group comparison and a program trial, in which the subjects are recruited according to a systematic allocation by order.

Since in the field of psychotherapy, "measure means affect," there is a built-in difficulty in building control groups (which are also committed to evaluation). For this reason, the proposed study combines a control group comparison.

Research population: The study will be carried out in the therapeutic settings of two psychiatric hospitals: the Shalvata Mental Health Center and the Geha Mental Health Center. The study population will include patients receiving therapeutic services in the ambulatory system of these centers (three clinics, the Shalvata Mental Health Center, one clinic, the Geha Mental Health Center). The study population includes patients with all the common mental disorders (adjustment disorders, anxiety, depression, personality disorders and somatomorphic disorders). The allocation between caregivers will be random in order, in a one-to-one ratio.

Research groups: The proposed study has two groups. Both groups include patients who are actively receiving psychotherapy on a weekly basis for at least three months to neutralize the effects of starting treatment. The first group will be under the usual treatment conditions (TAU); The second group will be exposed to a multidisciplinary therapeutic program that has a monitoring component and after two months an intervening component will be. In order to reduce the effect of the treated variables and the analysis of nested data, each therapist will introduce two patients into the study: one patient will be in the normal treatment condition (TAU) and the other under the monitoring and intervention program. In order to ensure randomization in this allocation, the clinic manager will determine the identity of the patients (i.e., each therapist will recruit two patients, and the allocation decision will be made anonymously by the clinic manager).

Inclusion criteria: Included are patients over the age of 18 years who have agreed to participate in the study, were found suitable for psychotherapeutic treatment and are treated with the attending clinician for at least two months. Patients who (due to cognitive impairment, language gaps, etc.) are not able to complete questionnaires with little help will not be included in the study. In order to minimize the effect of external variables, patients who, in the opinion of the clinician, are expected to undergo significant pharmacological changes (change in non-sleeping drugs or occasional sedatives) will not be inclusesd Population of caregivers: Experienced therapists from various therapeutic professions (including psychologists, social workers, psychiatrists, and other therapists who are graduates of psychotherapy training programs) will participate in the study. Only therapist who have a proven experience of at least 6 months in the clinic and manage at least four treatments at the beginning of the study will participate.

Data collection: Data collection will be carried out through computerized information systems (computerized medical records, by an application on a cellular device currently being developed as part of the project).

Research tools and variables: The primary outcome measure of the study is the OQ-45 (Lambert, M. J., Gregersen, A.T., Burlingame, G.M. (2004). The Outcome Questionnaire-45 The use of psychological testing for treatment planning and outcomes assessment: Volume 3: Instruments for adults (3rd ed) (pp. 191-234). Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers).

Methods of data analysis: Differences between groups will be examined using chi-squared tests (in categorical variables) or by independent T-tests and Mann-Whitney tests (non-categorical variables). Time differences will be analyzed by ANCOVA (repeated measures) and TSA (time series analysis). The sample size estimation is 68 patients.

Importance: Managed psychotherapeutic service has the potential to improve the clinical outcomes, and to increase the efficiency of the mental health services following the goals of the 2015 Mental Health Reform.

ELIGIBILITY:
Inclusion Criteria:

Included are patients over the age of 18 years who have agreed to participate in the study, were found suitable for psychotherapeutic treatment and are treated with the attending clinician for at least two months.

Exclusion Criteria:

Patients who (due to cognitive impairment, language gaps, etc.) are not able to complete questionnaires with little help will not be included in the study. In order to minimize the effect of external variables, patients who, in the opinion of the clinician, are expected to undergo significant pharmacological changes (change in non-sleeping drugs or occasional sedatives) will not be included

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in OQ45 | Initiation, Week 4, Week 7, Week 20
  The primary outcome measure of the study is the OQ-45 (Lambert, M. J., Gregersen, A.T., Burlingame, G.M. (2004). The Outcome Questionnaire-45 The use of psychological testing for treatment planning and outcomes assessment: Volume 3: Instruments for adults (3rd ed) (pp. 191-234). Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers).

IPD SHARING:
Plan to Share IPD: No